CLINICAL TRIAL: NCT00668434
Title: A Corticosteroid Taper for Acute Sciatica Treatment (The ACT FAST Study)
Brief Title: Effectiveness of Oral Prednisone in Improving Physical Functioning and Decreasing Pain in People With Sciatica
Acronym: ACT FAST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01AR053960 (NIH); R01AR053960 (NIH)
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Results first posted 2015-04-28 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Sciatica
Keywords: Back Pain; Leg Pain
MeSH Terms: conditions — Sciatica; Back Pain | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prednisone (Experimental): Participants will receive a 15-day tapering course of prednisone capsules.
  Interventions: Drug: Prednisone
- Placebo (Placebo Comparator): Participants will receive a 15-day course of placebo capsules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prednisone — For participants who weigh 50 kg or more, the prednisone dose will be 60 mg daily for 5 days, then 40 mg daily for 5 days, and then 20 mg daily for 5 days. For participants who weigh less than 50 kg, the dose will be 40 mg daily for 10 days, and then 20 mg daily for 5 days.
  Arms: Prednisone
Drug: Placebo — Placebo capsules will look the same as the study medication but will not contain active medicine.
  Arms: Placebo

SUMMARY:
Sciatica is a condition that causes a sharp, burning pain in the back, buttock, and leg. The condition is caused by injury to or compression of the sciatic nerve, which is located in the back of the leg. This study will determine the effectiveness of the steroid prednisone in decreasing pain and improving function in people with sciatica.

DETAILED DESCRIPTION:
Sciatica is most often caused by a herniated disc in the lumbar region of the back and results from inflammation of the nerve roots as they exit the spine. It is a very common cause of back and leg pain, loss of function, and inability to work. Although sciatica is common, the effectiveness of current treatments is limited. Epidural steroid injections (ESIs), which can reduce inflammation of the nerve roots, are commonly used to decrease sciatica pain and restore normal function in patients. The exact effectiveness of ESIs, however, is unknown. If inflammation, and not compression, is the main cause of sciatica, it is reasonable to consider giving the steroid orally rather than by injection. If oral steroids prove effective, patients and clinicians will have access to a simple, inexpensive therapy that can be prescribed by primary care physicians without delay. This study will determine the effectiveness of the oral steroid prednisone in decreasing pain and improving function in people with sciatica.

Participants in this study will attend a screening visit at which they will answer questions about their health to determine eligibility, undergo a neurologic exam, and have a plain lower spine x-ray. An MRI of the lower spine will be performed for those who meet clinical eligibility. Participants whose MRI shows that a disc has ruptured in a specific way will be randomly assigned to receive either a 15-day course of prednisone capsules or a 15-day course of placebo capsules. Participants will take their assigned study medications in addition to their usual pain medications.

At Week 3, participants will return for a follow-up visit during which they will answer questions about their pain and general health and wellness. Participants who are still having considerable pain will be offered an epidural steroid injection (ESI) as a part of the study. At Week 6, participants will be called at home for a telephone interview and again answer questions about their general health and wellness; this telephone call will last about 20 minutes. If they continue to have considerable pain, they will be offered a second ESI as part of the study.

At Week 12, an interviewer will phone participants to determine if their pain has decreased and whether they have been able to return to their normal activities. The telephone contact will last about 20 minutes. Additional information about their back problems will be obtained from their medical records and from Kaiser Permanente's computerized medical records on their use of health care and medicines for back problems. At Week 24, participants will attend an evaluation visit at the Spine Clinic to assess their progress and symptoms. At Week 52 (1 year from randomization), participants will undergo a final telephone interview.

ELIGIBILITY:
Inclusion Criteria:

* Seeks care at a Kaiser Permanente clinic spine care specialist at the San Jose, Redwood City, or Roseville site
* Complains of low back pain and functionally incapacitating leg pain extending below the knee with a nerve root distribution
* Score of at least 20 on the modified Oswestry Disability Index
* Appears, in the opinion of the study physician, to be very likely to have a herniated lumbar disc
* MRI study confirms a herniated disc consistent with the signs and symptoms

Exclusion Criteria:

* Onset of sciatica symptoms occurred more than 3 months before study entry
* Cauda equina syndrome
* Active cancer
* Acute spinal fracture
* Currently taking oral steroids
* Diabetes mellitus and taking insulin or glycohemoglobin greater than 10%
* Systolic blood pressure greater than 180 mm Hg or diastolic blood pressure greater than 110 mm Hg
* Pregnant or breastfeeding
* Active peptic ulcer disease
* History of intolerance to steroid therapy
* Bleeding diathesis or anticoagulant therapy
* Ongoing litigation or workers compensation claim for low back pain or sciatica
* Underwent previous lumbar surgery
* Received epidural steroid injection (ESI) within the 12 months before study entry
* Unable to read or speak English
* Progressive or severe motor loss

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2008-11; Primary Completion 2012-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harley Goldberg, DO, Principal Investigator — Kaiser Permanente San Jose Medical Center; Andrew L. Avins, MD, MPH, Principal Investigator — Kaiser Permanente Division of Research; William Firtch, MD, Principal Investigator — Kaiser Permanente Redwood City; Mark Tyburski, MD, Principal Investigator — Kaiser Permanente, Roseville
Locations (3):
- United States (3):
  - Kaiser Permanente Northern California, Redwood City, Redwood City, California
  - Kaiser Permanente, Roseville, California
  - Kaiser Permanente Northern California, San Jose, San Jose, California

REFERENCES:
- [Derived] Goldberg H, Firtch W, Tyburski M, Pressman A, Ackerson L, Hamilton L, Smith W, Carver R, Maratukulam A, Won LA, Carragee E, Avins AL. Oral steroids for acute radiculopathy due to a herniated lumbar disk: a randomized clinical trial. JAMA. 2015 May 19;313(19):1915-23. doi: 10.1001/jama.2015.4468. PMID 25988461

RESULTS

PARTICIPANT FLOW:
Period: Primary Outcome Time Point (3 Weeks)
Arm/Group | Prednisone | Placebo
Started | 181 (Baseline) | 88 (Baseline)
Completed | 179 | 88
Not Completed | 2 | 0
Period: Secondary Outcome Time Point (52 Weeks)
Arm/Group | Prednisone | Placebo
Started | 179 (Baseline) | 88 (Baseline)
Completed | 157 | 77
Not Completed | 22 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prednisone | Placebo | Total
Number analyzed (Participants) | 181 | 88 | 269
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (11.8) | 46.7 (12.6) | 46.0 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 37 | 120
  Male | 98 | 51 | 149
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 4 | 5
  Asian | 24 | 8 | 32
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 3 | 3 | 6
  White | 129 | 50 | 179
  More than one race | 10 | 9 | 19
  Unknown or Not Reported | 12 | 14 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 28 | 62
  Not Hispanic or Latino | 147 | 60 | 207
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 181 | 88 | 269

OUTCOME MEASURES:

1. Primary Outcome: Oswestry Disability Index, v2
Description: The Oswestry Disability Index, v2 is a back-pain-specific measure of disability and functional status. It is measured on a 0-to-100 scale, with higher numbers indicating greater disability.
Time Frame: Baseline, Week 3 follow-up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 179 | 88
units on a scale | -19.0 (1.4) | -13.3 (1.7)

2. Secondary Outcome: Pain Numerical Rating Scale
Description: Ordinal scale of average level of pain as perceived by the participant over the prior 3 days; measured on a 0-to-10 scale, with higher numbers indicating greater pain.
Time Frame: Baseline, Week 3 follow-up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 179 | 88
units on a scale | -3.0 (0.2) | -2.8 (0.3)

3. Secondary Outcome: Oswestry Disability Index, v2
Description: as for outcome 1
Time Frame: Baseline, Week 52 follow-up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 157 | 77
units on a scale | -37.8 (1.5) | -30.4 (2.2)

4. Secondary Outcome: Pain Numerical Rating Scale
Description: as for outcome 2
Time Frame: Baseline, Week 52 follow-up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 157 | 77
units on a scale | -5.2 (0.2) | -4.6 (0.3)

ADVERSE EVENTS:
Time Frame: Entire study period, up to 52 weeks
Arm/Group | Prednisone | Placebo
Serious Adverse Events (participants affected / at risk) | 3/181 | 2/88
Other Adverse Events (participants affected / at risk) | 143/181 | 63/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prednisone (N=181) | Placebo (N=88)
Partial nephrectomy (Renal and urinary disorders) | 0 (0) | 1 (1) — Resection of renal cell carcinoma found incidentally on study imaging
Deep venous thrombosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Upper GI bleed (Gastrointestinal disorders) | 0 (0) | 1 (1)
Appendectomy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prednisone (N=181) | Placebo (N=88)
Cardiovascular problem (Cardiac disorders) | 3 (4) | 0 (0)
Dermatologic problem (Skin and subcutaneous tissue disorders) | 18 (56) | 10 (27)
Ear or eye disorder (Ear and labyrinth disorders) | 0 (0) | 2 (6)
Gastrointestinal problem (Gastrointestinal disorders) | 41 (85) | 8 (32)
Genitourinary problem (Renal and urinary disorders) | 3 (8) | 2 (8)
Neurologic problem (Nervous system disorders) | 17 (62) | 14 (34)
Psychiatric disorder (Psychiatric disorders) | 47 (78) | 15 (36)
Pulmonary problem (Respiratory, thoracic and mediastinal disorders) | 1 (8) | 0 (0)
Kidney problem (Renal and urinary disorders) | 0 (0) | 1 (2)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 13 (45) | 11 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No